CLINICAL TRIAL: NCT03227419
Title: Abatacept Versus Tocilizumab by Subcutaneous Administration for the Treatment of Rheumatoid Arthritis in TNF Alpha Inhibitor Inadequate Responder Patients: A Randomized, Open-labeled, Superiority Trial
Brief Title: Abatacept vs Tocilizumab for the Treatment of RA in TNF Alpha Inhibitor Inadequate Responders
Acronym: SUNSTAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-P0055
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Abatacept

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, randomized, open-label, superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab Prefilled Syringe (Experimental): Market approval recommendations will be respected. Treatment should be started within 7 days of randomization.
  The treatment protocol has no specific provision for treatment adaptation. Treatment will be managed in compliance with the marketing approval recommendations and drug labeling described below.
  Interventions: Drug: Tocilizumab Prefilled Syringe
- Abatacept Prefilled Syringe (Experimental): Market approval recommendations will be respected. Treatment should be started within 7 days of randomization.
  The treatment protocol has no specific provision for treatment adaptation. Treatment will be managed in compliance with the marketing approval recommendations and drug labeling described below.
  Interventions: Drug: Abatacept Prefilled Syringe

INTERVENTIONS:
Drug: Tocilizumab Prefilled Syringe — Treatment arm: tocilizumab (RoActemra®):
  162 mg weekly a schema for therapeutic adaptation with injection intervals determined according to transaminase levels or blood cell counts (neutropenia, thrombopenia) as recommended by Roche-Chugaï (see table below).
  Other Names: RoActemra
  Arms: Tocilizumab Prefilled Syringe
Drug: Abatacept Prefilled Syringe — Treatment arm: abatacept (Orencia®)
  125 mg weekly after an initial dose of 500 mg (body weight <60kg), 750 mg (body weight between 60 and 100 kg), or 1000 mg (body weight >100 mg) 24 hours before the first subcutaneous injection.
  Other Names: Orencia
  Arms: Abatacept Prefilled Syringe

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatoid disease in France, affecting 0.3% of the general population. Without effective treatment, the persistent inflammation causes invalidating pain and joint destruction, leading to major functional disability.

Biological agents have been proposed for patients with RA who have the most severe form of the disease and that are inadequate responder patients to conventional synthetic Disease-modifying antirheumatic drugs (csDMARDs). TNF inhibitors (TNFi) are historically proposed as the first biological DAMRD for inadequate responder patients to csDMARDs. A diverse therapeutic arsenal has become available in recent years with the development of non-anti-TNFα drugs whose mechanisms of action are different from the classical TNFi. This new biotherapy class includes tocilizumab and abatacept, two drugs recently available for subcutaneous administration that enables ambulatory care for patients who would otherwise require repeated in-hospital care.

The role of these new treatments in the therapeutic strategy has been emphasized by studies that demonstrated their efficacy as first-line treatments. However, in clinical practice, TNFi remain the most common first-line treatment for the majority of patients, non-anti-TNFα biological agents being reserved for inadequate responder patients.

In second line, several studies have investigated therapeutic strategies for inadequate responder patients to TNFi. Current data suggest that it could be wise to change the therapeutic target after failure of a first-line treatment with TNFi.

Data about the comparative efficacy of different biologics proposed after failure of a first-line treatment with TNFi are in progress. Meta-analyses from registries and academic trials conducted in France and The Netherlands suggest that non-anti-TNFα agents would have equivalent or superior efficacy compared with a second TNFi. This finding suggests clinicians to switch for an alternate therapeutic target after failure of a first-line TNFi.

Data comparing different non-anti-TNFα biologics in inadequate responder patients to TNFi are scare. Industrial trials have demonstrated sustained biological efficacy of non-anti-TNFα biologics after failure of a TNFi. However, there is very little solid data on the direct comparison between them.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatoid disease in France, affecting 0.3% of the general population. Without effective treatment, the persistent inflammation causes invalidating pain and joint destruction, leading to major functional disability as well as progressive structural damage resulting in major joint deformity.

Biologic agents are taking on an increasingly important role in the management of patients with an inadequate response to conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs).

Biological DMARD (bDMARD) therapy consists in the use of monoclonal antibodies or fusion proteins, administered intravenously or subcutaneously. The earliest developed biologic agents have been available for more than 15 years. Tumor necrosis factor alpha (TNFα), a pro-inflammatory cytokine, was the first cytokine successfully targeted by a biologic agent for RA treatment. TNF inhibitors (TNFi) are historically proposed as the first bDAMRD for inadequate responder patients to csDMARDs. More recently non-anti-TNFα drugs have emerged, with other biological targets such as interleukin-6 receptor (tocilizumab) or B- (rituximab) and T-lymphocytes (abatacept) that are implicated in the inflammatory response. Initially administered strictly intravenously, these drugs are now available in formulations adapted to subcutaneous administration, which allows ambulatory care for patients who otherwise would require repeated in-hospital care.

National and international guidelines, especially those issued in 2013 by the European League Against Rheumatism (EULAR) and also in 2013 by the French Society of Rheumatology now recommend first-line treatment not only with TNFi but also with non-anti-TNFα biologic agents. However, in routine practice, most clinicians preferably prescribe TNFi for the first-line regimen, reserving non-anti-TNFα drugs to TNFi inadequate responder patients.

There is a growing body of research focusing on first-line biologic agents but there is very little solid data on the direct randomized comparison between them. Actually, all three of the published studies have systematically compared a non-anti-TNFα biomedication versus TNFi (one study with a blinded design and two open studies).

The therapeutic strategy that should be adapted after failure of a TNFi regimen has also been investigated. Those studies favor non-anti-TNF drugs over an alternate TNFi.

There is adequate evidence of the efficacy of the different non-anti-TNFα biologic agents versus placebo after TNFi failure. In other hands, industrial trials have not provided any comparative data between drugs. An academic trial from The Netherlands using medico-economic performance as the primary outcome found no difference in efficacy between abatacept and rituximab (a non-anti-TNFα drug administered exclusively intravenously) after failure of a TNFi. Meta-analyses using data from care networks have not reported any difference between different non-anti-TNFα drugs after failure of a TNFi.

Data from national registries have provided interesting complementary information since in everyday practice these agents are generally used after failure of at least one TNFi. The Danish registry thus suggests that the therapeutic response would be better with tocilizumab than with abatacept. This observation was confirmed by an analysis of French registries data presented at the American College of Rheumatology (ACR) congress in November 2016 showing that tocilizumab exhibits superiority for treatment persistence over 2 years. These results were fully in agreement with the findings of the French ROC trial comparing intravenous administration of a second anti-TNFα drug versus a non-anti-TNFα agent after failure of an anti-TNFα drug that suggested a superiority of tocilizumab over abatacept in the subgroup of patients given a non-anti-TNFα agent. A recent Bayesian network meta-analysis showed better efficacy in the non-anti-TNFα groups for ACR20 in patients who responded insufficiently to an anti-TNFα.

Subcutaneous formulations have been recently developed for both tocilizumab and abatacept. Subcutaneous administration is important because it enables ambulatory care for a substantial number of patients who to date are recurrently hospitalized in day-care units for their intravenous infusions. Excepting specific situations, the subcutaneous formulation will be favored for a large majority of patients because of economic as well as practical considerations. Phase III trials have demonstrated the equivalence of the intravenous versus subcutaneous routes of administration focusing on efficacy and tolerance. The subcutaneous formulation is now also available for routine administration of both tocilizumab and abatacept. Nevertheless, despite large-scale industrial trials on drug equivalence, data issuing from clinical practice suggest a potential difference in the behavior of these two formulations which needs to be explored. Rituximab is apart in the treatment strategy because of its exclusive intravenous administration at spaced intervals and because it is used for specific patient profiles (extra-articular involvement, history of neoplasia, rheumatoid factor (RF) and anti-citrullinated protein antibody (ACPA) positivity). There is no perspective for the development of a subcutaneous formulation of rituximab for RA patients. Furthermore, the routine treatment schedule for rituximab (one-time injections at a mean interval of 9 months) would compromise comparison, especially short-term comparison, with other subcutaneous treatments.

These findings illustrate the need for a new multicentric, prospective, randomized trial designed to demonstrate the superiority of tocilizumab over abatacept in patients exhibiting inadequate response to a first anti-TNFα. A direct comparison of subcutaneous formulation is the need for the promising route of administration for future ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* RA according to the ACR/EULAR 2010 criteria
* inadequate response to a subcutaneously administered first-line TNFi defined as moderate to high disease activity (DAS28-ESR>3.2 and CDAI>10) after at least 3 months of treatment with a TNFi
* beneficiary of the French National Health Insurance Fund
* signed informed consent form
* for women of childbearing age: effective contraception during treatment period with engagement to continue such contraception for 14 weeks after last administration

Exclusion Criteria:

* counter-indication for one or other of the two drugs under study
* prior failure of the TNFi due to intolerance
* receiving ≥15 mg/day prednisone for more than 4 weeks
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months of the Clinical Disease Activity Index (CDAI) | 6 months
  The CDAI is a composite score combining clinical items only: Tender 28-joint count, Swollen 28-joint count, Patient Global Disease Activity (PGA), Evaluator"s Global Disease Activity (EGA). This score provides a numerical assessment reflecting disease activity independently of cute phase reactants.
  It will be measured at baseline and 6 months after inclusion

SECONDARY OUTCOMES:
Change from baseline of the disease activity score | 3, 6 and 12 months
  DAS28-ESR and DAS28-CRP: the disease activity score (DAS) is a composite score providing a numerical assessment based on the tender and swollen joint counts, the PGA VAS and the selected acute phase reactant (ESR or CRP).
Change from baseline of the Clinical Disease Activity Index (CDAI) | 3 and 12 months
  The CDAI is a composite score combining clinical items only: Tender 28-joint count, Swollen 28-joint count, Patient Global Disease Activity (PGA), Evaluator"s Global Disease Activity (EGA). This score provides a numerical assessment reflecting disease activity independently of cute phase reactants.
Change from baseline of the SDAI | 3, 6 and 12 months
  the simple disease activity index (SDAI) is a composite score providing a numerical assessment based on the tender and swollen joint count, the PGAVAS, the EGA VAS, and CRP
Change from baseline in HAQ quality-of-life scores | 3, 6 and 12 months
Change from baseline in SF-36 quality-of-life scores | 3, 6 and 12 months
Change from baseline in disease self assessment | 3, 6 and 12 months
  FLARE-RA score
Change from baseline in Patient's Pain Assessment (PPA) | 3, 6 and 12 months
Change from baseline in PGA visual analogic scale (VAS) | 3, 6 and 12 months
Proportion of patients having achieved low disease activity | 3, 6 and 12 months
  Low disease activity (LDA) is defined as DAS28-ESR<3.2 (LDA-DAS28-ESR) and CDAI<10 (LDA-CDAI)
Proportion of patients in good or moderate EULAR therapeutic response | 3, 6 and 12 months
  Good or moderate EULAR therapeutic response is defined as at least 0.6-point reduction in DAS28-ESR and final DAS28-ESR<5.1
Proportion of patients achieving ACR20 response | 3, 6 and 12 months
  ACR20 response correspond to a 20% improvement in the following parameters: number of tender joints; number of swollen joints; 3/5 complementary items (PPA VAS, PGA VAS, EGA VAS, self-administered functional status questionnaire, acute phase reactant)
Proportion of patients achieving ACR50 response | 3, 6 and 12 months
  ACR50 responses correspond respectively to a 50% improvement in the following parameters: number of tender joints; number of swollen joints; 3/5 complementary items (PPA VAS, PGA VAS, EGA VAS, self-administered functional status questionnaire, acute phase reactant)
Proportion of patients achieving ACR70 response | 3, 6 and 12 months
  ACR70 response correspond respectively to a 70% improvement in the following parameters: number of tender joints; number of swollen joints; 3/5 complementary items (PPA VAS, PGA VAS, EGA VAS, self-administered functional status questionnaire, acute phase reactant)
Rates of treatment persistence | 3, 6 and 12 months
Rates of patients presenting at least one adverse events | 3, 6 and 12 months
Rates of treatment withdrawals for intolerance | 3, 6 and 12 months
Rates of treatment withdrawals for intolerance requiring in-hospital care | 3, 6 and 12 months
Rates of cardiovascular events | 3, 6 and 12 months
Rates of perturbation of the lipid profile | 3, 6 and 12 months
Rates of severe infection requiring in-hospital care | 3, 6 and 12 months
Rate of rescue medication use authorized by the protocol and treatment dose of patients achieving treatment persistence | 3, 6 and 12 months
Changes in joint US-Doppler synovitis and Doppler hyperemia grade of the hands and wrists | 6 months
Changes in Sharp score in hands, wrists and feet X-Ray | 12 months
Change in vascular endothelial growth factor (VEGF) levels | At 3 and 6 months
Changes in immunoglobulin (quantitative assay) | 6 months
Changes in interleukin-6 serum levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascart Tristan, MD, Principal Investigator — GHICL
Locations (26):
- France (26):
  - Hôpital Saint-Philibert, Lomme, Hauts-de-France
  - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - CH de Boulogne-sur-Mer, Boulogne-sur-Mer
  - Ch Cahors, Cahors
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble Hôpital Sud, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Lille, Lille
  - Clinique Infirmerie Protestante de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Lariboisière, Paris
  - CHU de Poitiers, Poitiers
  - CH René-Dubos, Pontoise
  - CHU de Reims, Reims
  - CHU Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU Saint-Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg
  - CHU de Tours, Tours
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascart T, Fautrel B, Gottenberg JE, Ducoulombier V, Richez C, Truchetet ME, Avouac J, Morel J, Basch A, Cormier G; SUNSTAR Study Group; CRI-IMIDIATE Network; Houvenagel E, Mariette X, Norberciak L. Abatacept versus tocilizumab for the treatment of rheumatoid arthritis in TNF inhibitor inadequate responders: study protocol of the SUNSTAR randomised controlled open-label superiority trial. BMJ Open. 2025 Jun 17;15(6):e098298. doi: 10.1136/bmjopen-2024-098298. PMID 40527572